CLINICAL TRIAL: NCT03174379
Title: A Pilot Study to Analyze the Effect of Acupuncture on Mobility And Quality of Life in Multiple Sclerosis
Brief Title: A Study to Analyze the Effect of Acupuncture on Mobility And Quality of Life in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-00440
Record Dates: First submitted 2017-05-31; First posted 2017-06-02 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Standard of Care; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Standard of Care (SOC) treatment will be based upon Traditional Chinese Medicine (TCM) interpretation of 4 phases of MS.
  Interventions: Procedure: Standard of Care with no acupuncture
- Treatment Group (Active Comparator): 60-minute treatment session twice a week for three weeks
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Standard of Care with no acupuncture — The control group will lie on a treatment table in the acupuncturist's office for the same amount of time that the treatment group did, but receive no acupuncture
  Arms: Control Group
Procedure: Acupuncture — The first set consists of core point selection, used in an MS Standard of Care (SOC). The second set of points will be individualized to the patient's needs as determined by the acupuncturist. SOC treatment will be based upon Traditional Chinese Medicine (TCM) interpretation of 4 phases of MS.
  Arms: Treatment Group

SUMMARY:
The purpose of this two-center study is to examine the effectiveness of acupuncture treatments in addressing mobility deficits, sensorimotor impairment, and quality of life (QOL) limitations in persons with Multiple Sclerosis (MS). It is hypothesized that acupuncture will result in an improvement in these limitations.

DETAILED DESCRIPTION:
This research study will examine the effects of acupuncture on various symptoms experienced by persons with MS. Persons with MS often use acupuncture as a way of controlling the symptoms of the disease. However, there is little research on whether or not acupuncture has any effect on MS symptoms related to movement. This study intends to look at the effects of acupuncture treatment on walking, balance, and mood in persons with MS.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MS
* ability to walk unaided for 6 minutes with or without assistive device

Exclusion Criteria:

* bleeding precautions
* trypanophobia
* inability to lie still for 30 minutes
* active cancer, current exacerbation, and history of previous acupuncture treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
fatigue severity scale | 14 Weeks
  The Fatigue Severity Scale (FSS) is a method of evaluating the impact of fatigue. The FSS is a short questionnaire that requires patient to rate level of fatigue.
Medical Outcomes Study Pain Effects Scale | 14 Weeks
  The MOS covers pain severity in terms of intensity, frequency, and duration while recording the impact on behaviours and moods. MOS contains twelve self report items on the severity of pain over the past four weeks and its effect on mood and behaviours
Gait measured by 6-minute walk test | 14 Weeks
  Assesses distance walked over 6 minutes as a sub-maximal test of aerobic capacity/endurance
Balance measured by 25-foot walk test | 14 Weeks
  The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-walk.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Siminovich-blok, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States